CLINICAL TRIAL: NCT01723579
Title: An Open-label, Multi-center Trial to Evaluate the Contraceptive Efficacy, Safety and Acceptability of a Monophasic Combined Oral Contraceptive (COC) Containing 2.5 mg Nomegestrol Acetate (NOMAC) and 1.5 mg Estradiol (E2) in Indian Women. Protocol MK-8175A-017-00
Brief Title: Efficacy and Safety of Oral NOMAC-E2 in Indian Women (P07057/MK-8175A-017)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P07057; MK-8175A-017 (Other: Merck)
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Contraception
MeSH Terms: interventions — nomegestrol acetate; Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NOMAC-E2 2.5 mg/1.5 mg (Experimental): Participants will receive combined oral contraceptive NOMAC-E2 2.5 mg/1.5 mg tablet for 13 consecutive 28-day cycles. Each 28-day cycle with consist of 24 active tablets and 4 placebo tablets taken at approximately the same time each day.
  Interventions: Drug: Nomegestrol acetate (NOMAC); Drug: Estradiol (E2)

INTERVENTIONS:
Drug: Nomegestrol acetate (NOMAC) — Oral tablet with daily release of 2.5 mg
Drug: Estradiol (E2) — Daily release of 1.5 mg

SUMMARY:
This study will investigate the efficacy and safety of the monophasic

combined oral contraceptive (COC) containing 2.5 mg NOMAC and 1.5 mg E2 in

healthy fertile Indian women.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active and at risk for pregnancy
* Of Indian descent, born in India, never emigrated out of India, with Indian

home address

* Body mass index (BMI) ≥17 and ≤35 kg/m^2

Exclusion Criteria:

* Presence or history of venous or arterial thrombotic/thromboembolic events

or cerebrovascular accident

* Presence or history of prodromi of a thrombosis
* History of migraine with focal neurological symptoms
* Diabetes mellitus with vascular involvement
* Presence of a severe or multiple risk factor(s) for venous or arterial

thrombosis

* Severe hypertension
* Severe dyslipoproteinemia
* Presence or history of pancreatitis associated with severe

hypertriglyceridemia

* Presence or history of severe hepatic disease
* Undiagnosed vaginal bleeding
* Known or suspected pregnancy
* Currently breastfeeding or breastfeeding within 2 months of starting

trial medication

- Investigational drug use or participation in another clinical trial within

2 months of signing Informed Consent Form for current trial

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Number of In-treatment Pregnancies | Day 1 of Treatment Cycle 1 Through Day 28 of Treatment Cycle 13, plus up to 2 additional days (Study Days 1-366)

SECONDARY OUTCOMES:
Number of Participants Experiencing an Adverse Event (AE) or Serious AE | "From Visit 1 up to 30 days after the last dose of study medication (up to Study Day 394).